CLINICAL TRIAL: NCT03045419
Title: Added Value of Gadoxetic Acid-enhanced Liver Magnetic Resonance Imaging for Diagnosis of Small (10-19 mm) or Atypical Hepatic Nodules at Contrast-enhanced Computed Tomography: A Prospective Study
Brief Title: Added Value of Gadoxetic Acid-enhanced Liver MRI
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Other Study IDs: SNUH-2009-5441
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Hcc; Diagnosis
Keywords: MRI; gadoxetic acid; CT
MeSH Terms: conditions — Carcinoma, Hepatocellular; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients group: * with small hepatic nodules (10-19mm) or atypical hepatic nodule (= or > 20mm) and high-risk group of HCC
  * scheduled for gadoxetic acid-enhanced liver MRI or liver nodule biopsy
  Interventions: Procedure: gadoxetic acid-enhanced liver MRI
- Living liver donor candidates: * living liver donor candidates without history of liver disease
  * schedule for gadoxetic acid-enhanced liver MRI as preoperative workup
  * only used for control of normal liver parenchymal enhancement on hepatobiliary phase
  Interventions: Procedure: gadoxetic acid-enhanced liver MRI

INTERVENTIONS:
Procedure: gadoxetic acid-enhanced liver MRI — liver MRI using a standard dose (0.025mmol/kg) of gadoxetic acid

SUMMARY:
It would be valuable to evaluate whether gadoxetic acid-enhanced liver MRI would provide additional value for characterizing atypical or small (1~2cm) hepatic nodules at CT and to reduce the necessity of biopsy in patients with high risk of HCC.

Therefore, the purpose of this study is to evaluate added value of gadoxetic acid-enhanced MRI for diagnosis of HCC in patients with small (10-19mm) or atypical hepatic nodules at CT.

DETAILED DESCRIPTION:
In terms of confirmative diagnosis, HCC is unique compared with other malignant tumors, as it can be diagnosed noninvasively based on its characteristic imaging features, that is, arterial hyperenhancement (washin) and hypoenhancement (washout) on portal or delayed phase at contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) using extracellular contrast media (ECCM). According to Liver Imaging Reporting and Data System (LI-RADS), hypointensity and isointensity on hepatobiliary phase (HBP) at gadoxetic acid-enhanced MRI are suggestive of malignancy and benignity, respectively, and those features are uniquely provided by only hepatocyte-specific contrast agent. However, these features are not included in diagnostic criteria because of its non-specificity, and indeed, gadoxetic acid-enhanced MRI is not yet included in AASLD and EASL guidelines as a diagnostic modality. If gadoxetic acid-enhanced MRI would provide better performance to diagnose HCC than CT, gadoxetic acid-enhanced MRI should be considered as a next step before biopsy in those small and/or atypical nodules to avoid potential diagnostic pitfall and morbidity, which is currently depending on physicians' decision. Thus, it would be valuable to evaluate whether gadoxetic acid-enhanced liver MRI would provide additional value for characterizing atypical or small (1~2cm) hepatic nodules at CT and to reduce the necessity of biopsy in patients with high risk of HCC.

Therefore, the purpose of this study is to evaluate added value of gadoxetic acid-enhanced MRI for diagnosis of HCC in patients with small (10-19mm) or atypical hepatic nodules at CT.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic hepatitis B or cirrhosis of any etiology
* signed informed consent AND
* being referred to radiology department for gadoxetic acid-enhanced MRI due to small nodule (10-19mm) at contrast-enhanced CT scan within 30 days as an radiofrequency ablation (RFA) work-up OR
* being referred to radiology department for percutaneous biopsy for atypical hepatic nodules (≥20mm) detected at contrast-enhanced CT within 30 days before biopsy

Exclusion Criteria:

* Any contraindication for MRI and MR contrast agent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients at a risk of HCC and had focal liver lesion at CT.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2009-12-29 (Actual); Primary Completion 2013-11-24 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
sensitivity to diagnose HCC, per-nodule base | 12 months after MRI
  sensitivity of HCC on CT and gadoxetic acid MRI, per-nodule base

SECONDARY OUTCOMES:
specificity to diagnose HCC, per-nodule base | 12 months after MRI
  specificity of HCC on CT and gadoxetic acid MRI, per-nodule base
sensitivity to diagnose HCC, per-patient base | 12 months after MRI
  sensitivity of HCC on CT and gadoxetic acid MRI, per-patient base
specificity to diagnose HCC, per-patient base | 12 months after MRI
  specificity of HCC on CT and gadoxetic acid MRI, per-patient base

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No